CLINICAL TRIAL: NCT00254085
Title: Multiple Substitution of First Phase Insulin Response With a Rapid Action Insuli Analogue in Patient With Newly Diagnosed Type 2 Diabtes.
Brief Title: Substitution of First Phase Insulin Response in Patient With Type 2 Diabetes.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2612-2368; KA 03092s
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-09

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabtes; Postprandial hyperglycemia; Insulin treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Insulin Aspart

INTERVENTIONS:
Drug: Insulin Aspart

SUMMARY:
The purpose of the project is to shown whether a little dose of a short acting insulin analogue given 3 time daily before the meals compared with placebo could normalise the increase in blood glucose after teh meals in diet treated Type 2 diabetic patients.

DETAILED DESCRIPTION:
Patients with Type 2 diabtes has a defect in the insulinsecretion combined with an increased insulin resistance. At an intravenously glucosestimulation, patients with Type 2 diabtes has a decresed first phase insulin response compared to healty peoples. Because the hyperglycemia after meal, observed i Type 2 diabetics patients, is related to the defect in the first phase insulin response it is our hypothesis that substitution of the first phase insulin response with a little dose of insulin could normalise the blood glucose after the meal.

20 patients with Type 2 diabetes will in a randomised, placebocontrolled, dobble-dummy study be included for three days treatment with Insulin aspart vs placebo. Primary endpoint is bloodglucose fluctuations monitored by a continously glucose monitor.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabtes according to the WHO criteria Fasting blood glucose >7 HbA1c between 6-9 Normal liver function Normal renal function

-

Exclusion Criteria:

Ongoing treatment with antidiabetic medicine Pregnancy and lactation -

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Blood glucose fluctuations

SECONDARY OUTCOMES:
number of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Gredal, MD, Principal Investigator — Gentofte University Hospital
Locations (1):
- Gentofte University Hospital, Hellerup, Hellerup, Denmark

REFERENCES:
- [Derived] Gredal C, Rosenfalck AM, Dejgaard A, Hilsted J. Targeting postprandial hyperglycaemia in patients with recently diagnosed type 2 diabetes with a fixed, weight-based dose of insulin Aspart. Scand J Clin Lab Invest. 2008;68(8):739-44. doi: 10.1080/00365510802207982. PMID 19016075